CLINICAL TRIAL: NCT05686642
Title: A Phase II Multicenter, Randomized, Double-blind, Placebo-controlled, Parallel-group Clinical Study to Evaluate the Safety and Efficacy of LT3001 in Subjects With Acute Ischemic Stroke (AIS)
Brief Title: Efficacy and Safety of LT3001 on Treating the Acute Ischemic Stroke
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Pharmaceuticals Holding Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SPH-LT3001-202
Record Dates: First submitted 2023-01-09; First posted 2023-01-17 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2025-04

CONDITIONS: Acute Ischemic Stroke
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- LT3001 Drug:high dose (Experimental)
  Interventions: Drug: LT3001 Drug:high dose
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- LT3001 Drug:low dose (Experimental)
  Interventions: Drug: LT3001 Drug:low dose

INTERVENTIONS:
Drug: LT3001 Drug:high dose — Administered by intravenous infusion.
  Arms: LT3001 Drug:high dose
Drug: Placebo — Administered by intravenous infusion.
  Arms: Placebo
Drug: LT3001 Drug:low dose — Administered by intravenous infusion.
  Arms: LT3001 Drug:low dose

SUMMARY:
This phase II clinical study is designed to evaluate the safety and efficacy of LT3001 in the treatment of acute ischemic stroke

ELIGIBILITY:
Inclusion Criteria:

1. Subjects aged between 18 and 80 years at screening;
2. Clinical diagnosis of acute ischemic stroke that causes evaluable neurological impairment; 3.4 points ≤ NIHSS score ≤ 25 points at randomization;

4.Subjects who are able to receive the investigational drug within 24 hours after the onset of stroke; 5.Female subjects of childbearing potential or male subjects whose sexual partner are women of childbearing potential have no pregnancy plan and voluntarily take effective contraceptive measures during the study period and for 3 months after the last dose; 6.All subjects sign the informed consent form by themselves or their guardians after receiving complete study information.

Exclusion Criteria:

1. Subjects have received or plan to receive endovascular treatment and/or intravenous thrombolytic therapy recommended by Chinese Guidelines for Diagnosis and Treatment of Acute Ischemic Stroke 2018 during this onset period;
2. Presence of disturbances of consciousness at screening and NIHSS 1a ≥ 2 points;
3. Neurological signs have improved rapidly and spontaneously at screening;
4. Subjects who have used or are using protocol-prohibited medications after the onset;
5. Subjects with pre-stroke disability;
6. Subjects with intracranial hemorrhagic diseases, tumor in brain parenchyma, arteriovenous malformation, aortic arch dissection, other central nervous system lesions that may increase the risk of hemorrhage, or imaging evidence for arterial aneurysm requiring treatment;
7. Massive infarction on imaging;
8. Patients who are unable to cooperate due to epileptic seizure at the onset of stroke or other concomitant mental disorders or are unwilling to cooperate;
9. Systolic blood pressure > 180 mmHg and/or diastolic blood pressure > 100 mmHg after active antihypertensive therapy;
10. Acute hemorrhage tendency;
11. Blood glucose level < 50 mg/dL or > 400 mg/dL;
12. Active visceral hemorrhage;
13. Lactating or pregnant subjects, or women of childbearing potential with positive pregnancy test results;
14. International normalized ratio > 1.7 or prothrombin time > 15 s;
15. Subjects with a history of serious hypersensitivity;
16. Subjects who experienced AIS, ICH, acute myocardial infarction or serious head trauma before screening;
17. Subjects who underwent any major surgery before screening;
18. Subjects with a history of active digestive ulcer before screening;
19. Subjects who experienced hemorrhagic disease before screening;
20. Subjects who underwent arterial puncture at the site not easy for hemostasis by compression before screening;
21. Serious hepatic impairment or serious renal insufficiency;
22. Subjects who have participated in another investigational study and used investigational product before screening;
23. Other conditions unsuitable for participation in this study determined by the Investigator.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2023-04-06 (Actual); Primary Completion 2025-12-10 (Estimated); Study Completion 2025-12-12 (Estimated)

PRIMARY OUTCOMES:
Incidence Adverse Events | Approximately 2 years
  Adverse event type, incidence, duration, correlation with study drug

SECONDARY OUTCOMES:
Proportion of subjects by mRS（Modified Rankin Scale） score (0 - 2) | Day 30 and Day 90 after the first dose
  Proportion of subjects by mRS score (0 - 2)
Proportion of subjects with an NIHSS（National Institute of Health stroke scale ） score of ≤ 1 point and/or with a decrease of ≥ 4 points from baseline in NIHSS score | Day 14 after the first dose
  Proportion of subjects with an NIHSS score of ≤ 1 point and/or with a decrease of ≥ 4 points from baseline in NIHSS score
Absolute change from baseline in NIHSS score | Day 3、Day 7、Day 14 and Day 30 after the first dose
  Absolute change from baseline in NIHSS score
Proportion of subjects with a BI（Barthel index） score of ≥ 95 points and ≥ 75 points | Day 30 and Day 90 after the first dose
  Proportion of subjects with a BI score of ≥ 95 points and ≥ 75 points

CONTACTS AND LOCATIONS:
Locations (28):
- China (28):
  - Beijing Luhe Hospital Capital Medical University, Beijing, Beijing Municipality
  - The First Affiliated Hospital of Jinan University, Guangzhou, Guangdong
  - Luoyang Third People's Hospital, Luoyang, He'nan
  - Harrison International Peace Hospital, Hengshui, Hebei
  - Daqing Oilfield General Hospital, Daqing, Heilongjiang
  - Zhongnan Hospital of Wuhan University, Wuhan, Hubei
  - The First Affiliated Hospital of Baotou Medical College, Baotou, Inner Mongolia
  - Inner Mongolia Baogang Hospital, Baotou, Inner Mongolia
  - Huai'an Second People's Hospital, Huai'an, Jiangsu
  - The Second Affiliated Hospital of Soochow University, Suzhou, Jiangsu
  - The Affiliated Hospital of Xuzhou Medical University, Xuzhou, Jiangsu
  - Pingxiang People's Hospital, Pingxiang, Jiangxi
  - The First Bethune Hospital of Jilin University, Changchun, Jilin
  - Beipiao Central Hospital, Chaoyang, Liaoning
  - Liaocheng People's Hospital, Liaocheng, Shandong
  - Yan'an University Xianyang Hospital, Xianyang, Shanxi
  - Xi'an Gaoxin Hospital, Xi’an, Shanxi
  - The Third Hospital of Mianyang, Mianyang, Sichuan
  - Zhejiang Hospital, Hangzhou, Zhejiang
  - Taizhou Municipal Hospital, Taizhou, Zhejiang
  - Taizhou First People's Hospital, Taizhou, Zhejiang
  - Beijing Tiantan Hospital, Capital Medical University, Beijing
  - Beijing Tsinghua Changgung Hospital, Beijing
  - Linfen Central Hospital, Linfen
  - Linfen People's Hospital, Linfen
  - Nanshi Hospital of Nanyang, Nanyang
  - Shanghai Pudong Hospital, Shanghai
  - Central People's Hospital of Zhanjiang, Zhanjiang